CLINICAL TRIAL: NCT03582176
Title: PrEvention of Posttraumatic Joint contractuRes With Ketotifen 2
Acronym: PERK2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Kevin Hildebrand, Professor Department of Surgery, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PERK2_KAH; CDMRP-OR160026 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2018-03-25; First posted 2018-07-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Elbow Fracture; Elbow Injury; Elbow Dislocation
Keywords: Acute elbow fractures and/or dislocations
MeSH Terms: conditions — Elbow Fractures; Elbow Injuries | interventions — Ketotifen

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double blinded multicenter trial with 3 parallel groups (Ketotifen 2 mg or 5 mg or lactose placebo twice daily orally for 6 weeks)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lactose Placebo (Placebo Comparator): Lactose Placebo by mouth twice per day
  Interventions: Drug: Lactose Placebo
- Ketotifen Fumarate - 2mg (Active Comparator): Ketotifen Fumarate 2 mg by mouth twice per day
  Interventions: Drug: Ketotifen Fumarate 2mg; Drug: Ketotifen Fumarate 5mg
- Ketotifen Fumarate - 5mg (Active Comparator): Ketotifen Fumarate 5 mg by mouth twice per day
  Interventions: Drug: Ketotifen Fumarate 2mg; Drug: Ketotifen Fumarate 5mg

INTERVENTIONS:
Drug: Lactose Placebo — One capsule by mouth twice per day
  Arms: Lactose Placebo
Drug: Ketotifen Fumarate 2mg — 2 mg tablets (over-encapsulated into one capsule) by mouth twice per day
  Arms: Ketotifen Fumarate - 2mg; Ketotifen Fumarate - 5mg
Drug: Ketotifen Fumarate 5mg — 5 mg tablets (over-encapsulated into one capsule) by mouth twice per day
  Arms: Ketotifen Fumarate - 2mg; Ketotifen Fumarate - 5mg

SUMMARY:
PrEvention of posttraumatic contractuRes with Ketotifen 2 (PERK 2) is a Phase III randomized, controlled, double blinded multicenter trial with 3 parallel groups (Ketotifen 2 mg or 5 mg or lactose placebo twice daily orally for 6 weeks) and a primary endpoint of elbow extension-flexion range of motion (ROM) arc at 12 weeks post-randomization.

DETAILED DESCRIPTION:
PrEvention of posttraumatic contractuRes with Ketotifen 2 (PERK2) is a Phase III randomized, controlled, double blinded multicenter trial with 3 parallel groups (Ketotifen 2 mg or 5 mg or lactose placebo twice daily orally for 6 weeks) and a primary endpoint of elbow extension-flexion range of motion (ROM) arc at 12 weeks post-randomization. The Research Hypothesis is that Ketotifen is superior to a lactose placebo in reducing joint contracture severity in adult participants with isolated elbow fractures or dislocations. The Primary Objective is to determine if Ketotifen given within 10 days of injury can reduce post-traumatic elbow joint contractures when compared to placebo. The Secondary Objectives are: 1) to ascertain the optimal dose of Ketotifen and 2) to compare adverse events in Ketotifen and placebo groups.

Inclusion criteria: age ≥ 18 years old and skeletally mature; distal humerus (AO/OTA type 13) and/or proximal ulna and/or proximal radius fractures (AO/OTA type 2U1/2R1) and/or elbow dislocations (open fractures with or without nerve injury may be included); injury ≤ 10 days; ability to give informed consent; able to comply with protocol and follow up; operative treatment of the elbow fracture or dislocation; participant has negative urine or blood serum pregnancy test.

Exclusion criteria: Pre-existing elbow contracture; elbow arthritis (osteoarthritis, inflammatory arthritis, or nonspecific monoarticular arthritis); inability to mobilize elbow within 21 days of injury; bilateral elbow injury; oral hypoglycemic medications; history of epilepsy; lactose intolerance; language or cognitive difficulties preventing completion of questionnaires; pregnancy; breast feeding; male or female unwilling to use 2 methods of contraception; total elbow replacement planned for treatment of fracture or dislocation; prior elbow injury or operation; concomitant musculoskeletal or visceral injuries preventing post-operative elbow therapy; severe renal and hepatic impairment.

Outcome Measures: Range of motion; Disability Arm, Shoulder, Hand; Oxford Elbow Score; Pain Catastrophizing Scale; standardized case report form; radiographic evaluation for fracture healing/non-union; and number of participants requiring reoperation for all elbow related causes, and post-traumatic joint contractures, 2 - 52 weeks post-randomization.

Safety Endpoints: The main safety endpoint for this study is the frequency of adverse events and serious adverse events, and radiographic assessment for non-union and heterotopic ossification (HO), 2 - 52 weeks post-randomization.

Ketotifen is the first and only agent demonstrating a significant decrease in contracture severity in preclinical trials that also has a wide safety profile. Ketotifen has been used in the treatment of chronic asthma for over 40 years in humans. Ketotifen is a medication that has anti-anaphylactic properties, due to the prevention of the synthesis and/or release of growth factors and mediators, as well as antihistamine affects due to H1 receptor antagonism. Post market surveillance has confirmed the safety of Ketotifen. A Phase II RCT comparing a single dose of Ketotifen (5 mg) to placebo in elbow fractures or dislocations in Calgary (ClinicalTrials.gov Identifier NCT01902017), demonstrated safety of Ketotifen and coupled with preclinical animal studies informed the need to increase the sample size, examine multiple doses, and narrow the study population to more severe injuries requiring an operation in the Phase III RCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old; skeletally mature with no growth plates in the elbow
* Distal humerus (AO/OTA type 13) and/or proximal ulna and/or proximal radius fractures (AO/OTA type 2U1 or 2R1) and/or elbow dislocations (open fractures with or without nerve injury may be included)
* Operative treatment of the elbow fracture or dislocation
* Injury ≤ 10 days
* Participant has a negative urine or blood serum pregnancy test

Exclusion Criteria:

* Pre-existing elbow contracture
* Elbow arthritis (osteoarthritis, inflammatory arthritis, or nonspecific monoarticular arthritis)
* Inability to mobilize elbow within 21 days of injury
* Bilateral elbow injury
* Concomitant musculoskeletal or visceral injuries preventing post-operative elbow therapy
* Oral hypoglycemic medications
* History of epilepsy
* Lactose intolerance
* Language or Cognitive difficulties preventing reliable completion of questionnaires
* Females who are pregnant or breast feeding
* Females of reproductive age or males unwilling to use 2 effective methods of contraception
* Severe renal impairment
* Severe hepatic impairment
* Prior elbow injury or operation
* Total elbow replacement planned for treatment of injury
* Unlikely to maintain follow up (no fixed address, plans to move out of town in the next year, states unable to comply with protocol)
* Unwilling or unable to provide written informed consent for trial participation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Elbow Extension-Flexion Arc of Motion | 12 weeks post-randomization
  The change in range of motion between baseline and 12 weeks post-randomization

SECONDARY OUTCOMES:
Range of Motion at other time points | 6 weeks, 24 weeks, 52 weeks
  Elbow extension-flexion arc of motion, forearm pronation-supination arc
Patient Reported Outcome Measures | Enrolment - 52 weeks
  Disability of the Arm, Shoulder and Hand (DASH) The upper extremity scoring scale DASH is a validated tool for disorders of the elbow with a range from 0 (least disability) to 100 (most disability). Ten is the average score in the general population and the minimal clinically important difference (MCID) is 10. DASH contains 30 questions asking participants about their ability to perform activities and their symptoms. Each question ranges from 1 (no difficulty) to 5 (unable). There is also optional work and sports/performing arts modules.
Patient Reported Outcome Measures | Enrolment - 52 weeks
  Oxford Elbow Score (OES). The OES is a 12-item questionnaire that is a valid measure of the outcome of surgery of the elbow in English (UK). It's 3 unidimensional domains include elbow function, pain, and social-psychological and the values range from 0 (greatest severity) to 100 (least severity). The OES has been used in trauma populations and its MCID is 10 for the elbow function domain and 18 for the pain and social-psychological domains.
Patient Reported Outcome Measures | Enrolment - 52 weeks
  Pain Catastrophizing Scale (PCS). The PCS is a 13-item instrument that can be completed in 5 minutes and requires a Grade 6 level of reading. For each question the participant has a choice from a range of 0 (not at all) to 4 (all the time). There are 3 subscale scores assessing rumination, magnification, and helplessness that are combined into an overall score. PCS total scores range from 0 - 52. Research at the University Centre for Research on Pain and Disability indicates that a total PCS score of 30 represents clinically relevant level of catastrophizing. It has been used in the assessment of injuries to the elbow, wrist, and hand where results are dependent on this behavior.
Radiographs | Enrolment - 52 weeks
  Radiographic evaluation for fracture healing and/or nonunion, and the number of participants requiring re-operation for contracture and also composite re-operation for all elbow related causes. This will be completed by a radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Hildebrand, MD, FRCSC, Principal Investigator — University of Calgary and Alberta Health Services
Locations (15):
- United States (3):
  - University of Maryland Medical Centre, Baltimore, Maryland
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Vermont Medical Center, Burlington, Vermont
- Canada (12):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - Royal Columbia Hospital, New Westminster, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Health Care London, London, Ontario
  - The Ottawa General Hospital, Ottawa, Ontario
  - The Ottawa Civic Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Ademola A, Hildebrand KA, Schneider PS, Mohtadi NGH, White NJ, Bosse MJ, Garven A, Walker REA, Sajobi TT. PrEvention of posttraumatic contractuRes with Ketotifen 2 (PERK 2) - protocol for a multicenter randomized clinical trial. BMC Musculoskelet Disord. 2020 Feb 24;21(1):123. doi: 10.1186/s12891-020-3139-2. PMID 32093652

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03582176/SAP_000.pdf